CLINICAL TRIAL: NCT03186365
Title: Efficacy of 8 Weeks Versus 12 Weeks of Elbasvir/Grazoprevir in Treatment-naïve Chronic Hepatitis C Genotype 1b Patients With Mild Fibrosis: an Open-label, Randomized, Active Control Trial (EGALITE)
Brief Title: 8 Weeks Versus 12 Weeks of Elbasvir/Grazoprevir in Treatment-naïve CHC With Mild Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISP-55740
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 8-week arm (Experimental): patients receiving 8 weeks of elbasvir 50 mg/grazoprevir (Zepatier Oral Product)100 mg daily
  Interventions: Drug: Zepatier Oral Product
- 12-week arm (Active Comparator): patients receiving 12 weeks of elbasvir 50 mg/grazoprevir 100 mg (Zepatier Oral Product) daily
  Interventions: Drug: Zepatier Oral Product

INTERVENTIONS:
Drug: Zepatier Oral Product — Grazoprevir, an HCV nonstructural protein 3/4A (NS3/4A) inhibitor 100 mg, plus elbasvir, an HCV NS5A inhibitor 50 mg fixed dose combination,Zepatier Oral Product, will be prescribed for 8-12 weeks
  Other Names: Zepatier

SUMMARY:
Grazoprevir plus elbasvir 12 to 16 weeks is now approved for chronic hepatitis C (CHC) genotype 1, 4, or 6 infection regardless liver disease severity. The current study aims to explore the efficacy and safety of 8-week grazoprevir/elbasvir in HCV-1b patients with mild liver fibrosis

DETAILED DESCRIPTION:
Grazoprevir, an HCV nonstructural protein 3/4A (NS3/4A) inhibitor 100 mg, plus elbasvir, an HCV NS5A inhibitor 50 mg fixed dose combination, Zepatier, achieved high SVR12 rates of > 95 % in treatment-naïve, experienced cirrhotic and non-cirrhotic patients with genotype 1, 4, or 6 infection. Zepatier, 12 to 16 weeks, was approved for the treatment of HCV genotype 1 and 4 in Taiwan in December, 2016. An SVR rate of 93 % was demonstrated in treatment-naive, non-cirrhotic (F0-F3) GT1b-infected patients who received 8 weeks of grazoprevir/elbasvir with or without ribavirin in the pooled analysis of C-WORTHY (PN035) and C-EDGE treatment-naive (PN060) trials. Furthermore, truncated treatment period of 8-week grazoprevir/elbasvir could achieve an even higher SVR rate at > 98% for naive HCV G1b patients with mild fibrosis (Fibrosis score 0-2). The study aims to evaluate the efficacy of 8-week regimen with grazoprevir/elbasvir on naïve, HCV G1b patients with mild fibrosis by a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve, HCV genotype 1b patients
* History of chronic HCV infection > 6 months
* Aged at least 20 years
* HCV RNA of 10,000 IU/mL or greater
* Fibroscan examination < 9.5 Kpa
* Negative serum or urine pregnancy test result (sensitivity of 25 mIU or better) for women with childbearing potential within the 24-hour period before the first dose of study drugs
* Female patients with childbearing potential must agree to use two reliable forms of effective non-hormonal contraception (i.e., condoms, cervical barriers, intrauterine device, spermicides, or sponge), at least 1 of which must be a physical barrier method, during treatment till end of follow up.
* A hormonal contraception (in lieu of non-hormonal) plus a physical barrier method can be used after end of treatment. All men with female partners of childbearing potential must use two reliable forms of effective contraception (combined) during treatment and till end of follow up
* Ability to participate and willingness to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

* Prior experience of IFN or direct antiviral agents (DAA)
* Hepatitis B virus or HIV co-infection.
* Patients with experience of ascites, esophageal varices, or other evidence of hepatic decompensation, and/or hepatocellular carcinoma.
* History of organ transplantation, except cornea transplantation.
* Hemoglobulin concentration < 11 mg/dl
* Platelet count < 75,000/mm3
* Albumin < 3 mg/dL
* History of active malignancy within the last 5 years, with the exception of localized or in situ carcinoma (e.g., basal or squamous cell carcinoma of the skin)
* Poorly controlled diabetes (Hemoglobin A1c value ≥ 8.5%) and endocrine condition.
* Total bilirubin >2 mg/dL, unless subject has a documented history of Gilbert's disease.
* Pregnant or lactating women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
the rate of subjects with undetectable HCV RNA 12 weeks post end-of-treatment | through study completion, an average of 5.5 months
  to determine the treatment efficacy (sustained virological response 12 weeks after treatment, SVR12) of 8 weeks of grazoprevir/elbasvir for naïve HCV G1b patients with mild fibrosis, compared to the SVR12 of a universal 12-week grazoprevir/elbasvir for naïve HCV G1b patients with mild fibrosis (Fibrosis score 0-2

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, MD., PhD., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CF, Hung CH, Cheng PN, Bair MJ, Huang YH, Kao JH, Hsu SJ, Lee PL, Chen JJ, Chien RN, Peng CY, Lin CY, Hsieh TY, Cheng CH, Dai CY, Huang JF, Chuang WL, Yu ML. An Open-Label, Randomized, Active-Controlled Trial of 8 Versus 12 Weeks of Elbasvir/Grazoprevir for Treatment-Naive Patients With Chronic Hepatitis C Genotype 1b Infection and Mild Fibrosis (EGALITE Study): Impact of Baseline Viral Loads and NS5A Resistance-Associated Substitutions. J Infect Dis. 2019 Jul 19;220(4):557-566. doi: 10.1093/infdis/jiz154. PMID 30957170